CLINICAL TRIAL: NCT01511848
Title: A Prospective Randomized Comparative Study of Efficacy and Safety of Combined Deferiprone (DFP) and Deferasirox Versus DFP and Desferrioxamine (DFO) Therapy in Diseases With Severe Iron Overload
Brief Title: Study Of Efficacy,Safety of Combined Deferasirox and Deferiprone Versus Combined Deferiprone and Desferal In Conditions of Iron Overload
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, professour of pediatrics, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AinShamsU
Record Dates: First submitted 2012-01-06; First posted 2012-01-19 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Beta-thalassemia Major; Sickle Cell Disease; Iron Hemosiderosis
Keywords: Iron chelation; Iron balance; Secondary iron overload; deferoxamine; deferasirox; Deferiprone; 1- Beta-thalassemia major patients;; Patients with high iron stores; Serum ferritin consistently > 2500 mcg/l and or increasing trend over previous 12 months; Liver iron >14 mg/g dry weight- by R2 MRI; 2- Sickle cell disease; 3- Other causes of transfusional iron hemosiderosis
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell | interventions — Isoflurophate; Deferiprone; Deferasirox; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm 1 (Active Comparator): 30 Patients will be treated with combined DFP and deferasirox.
  Interventions: Drug: DFP (ferriprox) and deferasirox (ICL 670)
- arm 2 (Active Comparator): Patients will be treated for 6 days with a combination of deferoxamine and DFP
  Interventions: Drug: DFP, DFO

INTERVENTIONS:
Drug: DFP (ferriprox) and deferasirox (ICL 670) — Drug: Ferriprox It will be given orally in the morning Other Name: DFP Initial dose 25/mg/kg 3 times/d (better tolerated if started and then built up over 4 weeks).
  Dose may be increased up to 100mg/kg/day guided by serum ferritin. Agranulocytosis risk 1-2%. Monitor TLC and granulocytic count / 2weeks. Patients need to be continually educated about this risk, know that they must stop DFP if they have a fever or infection.
  Drug: Deferasirox will be orally administered at a dose of 20 mg/kg once daily at evening for 5 days.
  Other Name: ICL670
  Arms: arm 1
Drug: DFP, DFO — Drug: Deferoxamine It will be administered subcutaneously over 8 hours for 5 days at a dose of 40 mg/kg.
  Other Name: Desferal, DFO Drug: DFP DFP: will be orally administered at a dose of 75mg/kg orally in 3 divided doses for 7 days
  Arms: arm 2

SUMMARY:
Interventional Allocation: Randomized Endpoint Classification: Safety/Efficacy Study of combined chelation therapy Masking: Open Label Primary Purpose: Treatment of transfusional iron overload

Primary Outcome Measures:

• The primary outcome measure is to assess efficacy in lowering serum ferritin level(the change in serum ferritin compared to baseline) with combining DFP and deferasirox compared to combined DFP and DFO in conditions with severe chronic iron overload; showing an up-trend of SF over previous 12 months on single chelator.

Secondary Outcome Measures:

• The secondary outcome measure is to determine the number of patients who will develop adverse events in order to assess safety upon administering the drugs in combination (DFP and DFX) compared to the combination of DFO and DFP.

DETAILED DESCRIPTION:
Study population:

1. Beta-thalassemia major patients; Patients with high iron stores Serum ferritin consistently > 2500 mcg/l and or increasing trend over previous 12 months Liver iron >14 mg/g dry weight- by R2 MRI
2. Other causes of transfusional hemosiderosis

Estimated Enrollment: 30 patients in each arm Study Start Date: January 1st ; 2011 enrollment period 8 weeks Estimated Study Completion Date: End of February 1212

Arms Assigned Interventions

Arm 1: Patients will be treated with combined DFP and deferasirox. Drug: Ferriprox It will be given orally in the morning Other Name: DFP Initial dose 25/mg/kg in 3 divided doses (better tolerated if started and then built up over 4 weeks).

Dose may be increased up to 100mg/kg/day guided by serum ferritin. Agranulocytosis risk 1-2%. Monitor TLC and granulocytic count / 2weeks. Patients need to be continually educated about this risk, know that they must stop DFP if they have a fever or infection.

Drug: Deferasirox will be orally administered at a dose of 20 mg/kg once daily at evening for 5 days.

Other Name: ICL670 Arm 2: Patients will be treated for 6 days with a combination of deferoxamine and DFP.

Interventions:

* Drug: Deferoxamine
* Drug: DFP Drug: Deferoxamine Deferoxamine will be administered subcutaneously over 8 hours for 5 days at a dose of 40 mg/kg.

Other Name: Desferal, DFO Drug: DFP DFP: will be orally administered at a dose of 75mg/kg orally in 3 divided doses for 7 days

Eligibility Ages Eligible for Study : 6 to 18Years Genders Eligible for Study: Both

Inclusion Criteria:

* Subjects with transfusional iron overload after Approval of Ethical committee giving written informed consent.
* Subjects must have a serum ferritin greater than >2500 ng/mL, a platelet count greater than 100,000/mm3, and a serum creatinine within the normal range.
* A woman of childbearing potential must have a negative serum pregnancy test at screening. She must use a medically acceptable form of birth control during the study and for 1 month afterward.
* The subjects must also have a level of understanding and willingness to cooperate with the confinement and procedures described in the consent form and scheduled by the study site. In addition, he/she must be able to provide voluntary written informed consent.

Exclusion Criteria:

* Subjects with a past history of agranulocytosis, history of clinically significant gastrointestinal, renal, hepatic ALT > 10 times high normal, OR > 50% increase of serum creatinine from basal value, pulmonary or cardiovascular disease. Patients with a history of tuberculosis, epilepsy, psychosis, glaucoma or any other condition, which in the opinion of the investigators, would jeopardize the safety of the subject or impact the validity of the study results.
* Subjects with HIV positive or have active HCV.
* A history of serious immunologic hypersensitivity to any medication, such as prophylaxis or angioedema.
* Participation in a previous investigational drug study within the 30 days preceding screening..
* Women who are pregnant, or breast-feeding.
* Current alcohol or drug abuse.
* An inability to adhere to the designated procedures and restrictions of this protocol.
* Subjects receiving warfarin, digoxin, or anti-arrhythmic or anti-seizure medications.
* Subjects with a known allergy to Exjade or DFP that prevents chronic administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with transfusional iron overload secondary to thalassemia major , sickle cell disease showing up-trend in SF aged 6 Years or older, may participate after Approval of Ethical committee giving written informed consent.
* Subjects must have a serum ferritin greater than >2500 ng/mL, a platelet count greater than 100,000/mm3, and a serum creatinine within the normal range.
* A woman of childbearing potential must have a negative serum pregnancy test at screening. She must use a medically acceptable form of birth control during the study and for 1 month afterward.
* The subjects must also have a level of understanding and willingness to cooperate with the confinement and procedures described in the consent form and scheduled by the study site. In addition, he/she must be able to provide voluntary written informed consent.

Exclusion Criteria:

* Subjects with a past history of agranulocytosis, history of clinically significant gastrointestinal, renal, hepatic ALT > 10 times high normal, OR > 50% increase of serum creatinine from basal value, pulmonary or cardiovascular disease. Patients with a history of tuberculosis, epilepsy, psychosis, glaucoma or any other condition, which in the opinion of the investigators, would jeopardize the safety of the subject or impact the validity of the study results.
* Subjects with HIV positive or have active HCV.
* A history of serious immunologic hypersensitivity to any medication, such as anaphylaxis or angioedema.
* Participation in a previous investigational drug study within the 30 days preceding screening..
* Women who are pregnant, or breast-feeding.
* Current alcohol or drug abuse.
* An inability to adhere to the designated procedures and restrictions of this protocol.
* Subjects receiving warfarin, digoxin, or anti-arrhythmic or anti-seizure medications.
* Subjects with a known allergy to Exjade or DFP that prevents chronic administration.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
to assess efficacy of combining DFP and deferasirox compared to combined DFP and DFO in decreasing the serum ferritin level in conditions with severe chronic iron overload. | 12 months
  • The primary outcome measure is to measure the change in serum ferritin level from baseline in the 2 combination therapy.

SECONDARY OUTCOMES:
to determine the safety upon administering the drugs in combination (DFP and DFX) compared to the combination of DFO and DFP. | 12 months
  • The secondary outcome measure is to determine the number of patients who will develop adverse reactions upon administering the drugs in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen S. Elalfy, professour, Principal Investigator — Ain Shams University
Locations (1):
- Pediatric Hematology clinic, Ain Shams University, Cairo, Egypt

REFERENCES:
- [Derived] Elalfy MS, Adly AM, Wali Y, Tony S, Samir A, Elhenawy YI. Efficacy and safety of a novel combination of two oral chelators deferasirox/deferiprone over deferoxamine/deferiprone in severely iron overloaded young beta thalassemia major patients. Eur J Haematol. 2015 Nov;95(5):411-20. doi: 10.1111/ejh.12507. Epub 2015 Mar 27. PMID 25600572